CLINICAL TRIAL: NCT06940661
Title: Obinutuzumab for Remission Induction in Patients With Relapsing PR3-ANCA Granulomatosis With Polyangiitis (Wegener's). Phase 2 Prospective, Open-label Study
Brief Title: Obinutuzumab for Remission Induction in Patients With Relapsing PR3-ANCA Granulomatosis With Polyangiitis
Acronym: OBI-WAN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP211000; 2022-501557-36 (EudraCT Number)
Record Dates: First submitted 2025-03-14; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Granulomatosis With Polyangiitis
Keywords: Relapsing PR3-ANCA granulomatosis with polyangiitis; Obinutuzumab
MeSH Terms: conditions — Granulomatosis with Polyangiitis | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Obinutuzumab — Patient will receive 1000 milligrams intravenous (IV) infusion on week 0, week 2, week 24 and week 26.
  Patients will receive the same standardized glucocorticoid tapering schedule (prescribe as a standard of care management and considered as auxiliary medicinal product)
  Premedication for obinutuzumab infusion related reactions (considered as auxiliary medicinal products) :
  * 100 mg methylpredinisolone
  * 1000 mg paracetamol
  * 5 mg dexchlorpheniramine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of obinutuzumab to induce clinical and serological remission in patients with relapsing PR3-ANCA granulomatosis with polyangiitis.

DETAILED DESCRIPTION:
Systemic vasculitides are rare inflammatory diseases of blood vessels, among which anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitides (AAV) are one of the most severe forms with life-threatening manifestations. In patients with AAV, the most important questions are how to achieve a long-term remission and prevent a relapse most effectively.

The pivotal RAVE trial showed that rituximab therapy was not inferior to daily cyclophosphamide treatment for induction of remission in AAV; and could be superior than cyclophoshamide in proteinase 3 (PR3)-ANCA patients. The MAINRITSAN trial, conducted by our group (Groupe Français d'Etude des Vascularites), has then demonstrated that more AAV patients had sustained remission with rituximab than with azathioprine.

However, despite its ability to induce and maintain remission, rituximab is associated with the occurrence of relapse after discontinuation in up to 50% of patients at 5-years in PR3-ANCA patients. Data strongly suggest that achieving clinical and serological remission (i.e. a BVAS (Birmingham Vasculitis Activity Score) of 0 and a negativation of ANCA) and longer B-cell depletion could be major goals to achieve in PR3-ANCA granulomatosis with polyangiitis to decrease the risk of relapse.

Obinutuzumab is a humanized type 2 antibody targeted against CD20. In preclinical studies, obinutuzumab showed superior efficacy, as compared with rituximab. In clinical studies, obinutuzumab was shown to be superior to rituximab in patients with chronic lymphocytic leukemia and follicular lymphoma, and met its primary and secondary endpoints in lupus nephritis.

The OBI-WAN study aims to evaluate the efficacy and safety of obinutuzumab to induce clinical and serological remission in patients with relapsing PR3-ANCA granulomatosis with polyangiitis. We hypothesize that obinutuzumab would induce higher remission rates and subsequent longer B-cell depletion compared to what is described for rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged of 18 years or older,
* Patients with relapsing granulomatosis with polyangiitis positive for PR3-ANCA (at initial diagnosis or during follow-up), according to the ACR/EULAR 2022 classification criteria, and/or the 2012 revised Chapel Hill Consensus Conference definition.
* Patients with an active disease defined as a Birmingham Vasculitis Activity Score (BVAS) ≥ 3,
* Patients within the first 21 days following initiation/increase of glucocorticoids at a dose ≤1 mg/kg/day (pulses of methylprednisolone before oral glucocorticoid therapy are authorized)
* Patient able to give written informed consent prior to participation in the study, - Affiliation with a mode of social security (profit or being entitled).

Exclusion Criteria

* Patients with MPO-positive AAV, or other vasculitis, defined by the ACR criteria and/or the Chapel Hill Consensus Conference,
* Patients with vasculitis in remission of the disease defined as a BVAS < 3,
* Patients with a newly-diagnosis of GPA
* Patients treated with rituximab within the last 6 months before inclusion
* Patients treated with cyclophosphamide within the last 6 months before inclusion
* Patients with severe cardiac failure defined as class IV in New York Heart Association
* Subject known to be seropositive for human immunodeficiency virus (HIV), hepatitis B (included history of previous infection) or hepatitis C
* Patients with active cancer or recent cancer (< 5 years), except basocellular carcinoma and prostatic cancer of low activity controlled by hormonal treatment,
* Patients with hypersensitivity to a monoclonal antibody or biologic agent,
* Patients with hypersensitivity to obinutuzumab or to its excipients
* Contra-indications to auxiliary medicinal products (methylprednisolone, paracetamol, prednisone, dexchlorpheniramine)
* Patients with other uncontrolled diseases, including drug or alcohol abuse, active infections or antecedents of chronic or recurrent infections, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol,
* Patients suspected not to be observant to the proposed treatments,
* Pregnant women and lactation. All women of childbearing potential (WOCBP) are required to have a negative pregnancy test (blood or urine) before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using an effective method of birth control from the date of consent through the end of the study, and at least 18 months after stopping obinutuzumab such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner,
* Men who refuse to use effective method of contraception (condom) from the date of consent through the end of the study and at least 18 months after stopping obinutuzumab (unless permanently sterile by bilateral orchidectomy or vasectomy),
* Patient participating in another investigational therapeutic study
* Protected adults (including individual under legal guardianship by court order or curatorship) or adults deprived of liberty
* Patients unable to give written informed consent prior to participation in the study.
* Patients with severe liver insufficiency (prothrombin time <50% and total bilirubin >50 micrmol/L)) or pulmonary insufficiency requiring nasal oxygen,
* Patients with an active infection or a history of chronic or recurrent infections
* Vaccination with live virus vaccines in the 4 weeks before study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients who achieved clinical and serological remission at week 24 (month 6) | week 24
  The percentage of patients who achieved clinical and serological remission at week 24 (month 6), defined by:
  * a BVAS of 0,
  * a negativation of PR3-ANCA,
  * and successful completion of the prednisone taper

SECONDARY OUTCOMES:
Proportion of participants experiencing adverse events and severe adverse events | Week 24 and 52
  The number of adverse events, expressed as adverse events according to the CTCAE toxicity grading system per patient-year at week 24 and 52 for the following adverse events combined: death (all causes), grade 2 or higher leukopenia or thrombocytopenia, grade 3 or higher infections, haemorrhagic cystitis, malignancies, venous thromboembolic events, hospitalization resulting either from the disease or from a complication due to the study treatment, infusion reactions (within 24 hours of infusion) that result in the cessation of further infusions,
Number and causes of deaths | Week 52
  Number and causes of deaths
Proportion of disease flares, including minor and major relapses | Week 52
  Proportion of participants who had vasculitis relapses (BVAS > 0), including minor and major relapses over the 12 months study periodCD19
Proportion of participants who remain with a BVAS of 0 during the treatment period with prednisone at a dose of less than 10 mg per day | Treatment period
  BVAS, prednisone dose
The time to B-cell repopulation defined by detectable CD19+ B cells in peripheral blood over the 12 months study period | Week 24 and 52
  CD19+ rate
The patient-reported outcomes (PRO) including HAQ and SF-36, patient-reported disease activity at week 24 and 52 | Week 24 and 52
  HAQ and SF-36 questionnaires
The Vasculitis Damage Index at week 24 and 52 | Week 24 and 52
  Vasculitis Damage Index (VDI)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PUECHAL, PhD, Study Director — Hôpital Cochin, Assistance Publique-Hôpitaux de Paris - Service de Médecine Interne, Centre de référence " Maladies systémiques et autoimmunes rares, en particulier Vascularites nécrosantes et Sclérodermies systémiques "
Locations (1):
- Service de Médecine Interne, Centre de reference "Maladies systémiques et autoimmunes rares, en particulier Vascularites nécrosantes et Sclérodermies systémiques", Paris, France